CLINICAL TRIAL: NCT06866496
Title: Disease and Outcomes in Alcohol Related Liver Cirrhosis - A Prospective Cohort Study of Optimized Remission
Brief Title: Optimized Remission in Alcohol-related Liver Cirrhosis
Acronym: Pro-ALC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Principal Investigator, Nina Kimer, Medical Specialist, Associate Professor, Copenhagen University Hospital, Hvidovre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-24053649; H-2024-16976 (Other: Scientitic Ethics Committee Capital Region of Denmark)
Record Dates: First submitted 2025-02-26; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-02

CONDITIONS: Cirrhosis of the Liver; Alcoholic Cirrhosis
Keywords: cirrhosis; ArLD
MeSH Terms: conditions — Fibrosis; Liver Cirrhosis, Alcoholic | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): Standard of care for liver cirrhosis, including treatment of alcohol use disorder.
  Interventions: Behavioral: Motivational interviews; Other: Standard of Care (SOC)

INTERVENTIONS:
Behavioral: Motivational interviews — Three short and structured motivational enhancement interviews to aid alcohol cessation.
Other: Standard of Care (SOC) — Standard of care including medical treatment of decompensation, nutrition support, medical treatment of alcohol withdrawal symptoms and craving

SUMMARY:
The incidence of liver cirrhosis is increased fivefold for men and tripled for women in the last forty years.

The clinical course of liver cirrhosis includes complications of ascites, hepatic encephalopathy, variceal bleeding, kidney dysfunction, and infections that markedly worsen prognosis. These complications are driven by the development of portal hypertension in the liver. This progression to the 'decompensated' stage is considered a hallmark in the disease course, as the decompensation is associated with a markedly increased risk of further complications and death.

Increasing evidence indicate that active measures of treatment of the underlying cause of liver disease and removal of the toxic agents causing cirrhosis may slow disease progression or even induce regression of cirrhosis. This concept is described as hepatic recompensation.

There is a need for clinical studies investigating novel biomarkers with the capability to predict and monitor improvement in alcohol related liver cirrhosis, Between 75% and 80% of patients with liver cirrhosis in Denmark have or have had a harmful use of alcohol.

Alcohol related liver disease (ArLD) has a major impact on patients' health and lives, and there is an unmet need to investigate treatment options that not only relieves complications, but also address the underlying pathways of alcohol related liver disease, also in severe stages of alcohol related cirrhosis (ALC). Factors such as BMI, female gender and mild portal hypertension are known to be associated with an increased likelihood of recompensation. Additional factors of genetic activation and molecular biomarkers from the proteome and lipidome have only attracted minor attention, and the impact of treating the drivers of decompensation, portal hypertension and alcohol use, and their impact on the natural cause of disease, have not been addressed.

The molecular pathophysiology of ArLD is incompletely understood. Characterization of the proteome dynamics across the spectrum of ALD could provide new insights into disease mechanisms of both progression and remission of disease.

Several markers of inflammation and cytokines are involved in driving decompensation and has the potential to predict the risk of early death. It is unknown whether such markers can predict remission and recompensation in ALC and AH. Prospective studies investigating the associations between biomarkers of metabolism and prognosis, monitoring and efficacy og treatment in ALC are missing.

The overall objective of the present study is to investigate the molecular profile and pathways in persons with ALD to support personalized monitoring and follow-up in liver cirrhosis.

The study is an incidence cohort in which patients will be followed from diagnosis to death or withdrawal from the cohort. We will seek to include patients consecutively within three months of diagnosis.

All patients with a debut of alcohol related liver cirrhosis during admission regardless of the reason for admission, are eligible for inclusion.

All participants in this study will be offered the standard of care treatment. Alcohol cessation intervention including medical treatment of withdrawal symptoms and craving, referral to municipal offers of alcohol treatment, and motivational interviews is part of the treatment.

The study will contribute to a better characterization of advanced liver disease related to alcohol and contribute to an improved future organization of treatment- and rehabilitation offers to patients with liver disease. thorough characterization and consecutive inclusion will enhance our understanding on the incidence, prevalence and impact of ALC in the population, as well as the utilization of health care resources allocated to its treatment.

A deeper insight into the molecular mechanisms of liver progression and remission will, in combination with clinical data, support our ability to predict outcomes in cirrhosis, facilitate personalized monitoring aiming at providing the right treatment for the right patient at the right time.

DETAILED DESCRIPTION:
In Denmark the incidence of liver cirrhosis is increased fivefold for men and tripled for women in the last forty years. In 2008 approximately 15,000 people were diagnosed with liver cirrhosis. Patients who are readmitted to the hospital have a higher 90-day mortality than those who avoid readmission.

The clinical course of liver cirrhosis includes complications of ascites, hepatic encephalopathy, variceal bleeding, kidney dysfunction, and infections with repeated admissions to hospital that markedly worsen prognosis. These complications are driven by the development of portal hypertension in the liver. This progression to the 'decompensated' stage is considered a hallmark in the disease course, as the decompensation is associated with a markedly increased risk of further complications and death.

Several clinical studies have sought to find medical remedies that prevent complications related to portal hypertension or slow down further progression in cirrhosis. Yet, increasing evidence indicate that active measures of treatment of the underlying cause of liver disease and removal of the toxic agents causing cirrhosis may slow disease progression or even induce regression of cirrhosis. This concept is described as hepatic recompensation.

Clinical and biochemical features such as BMI and albumin levels may be linked to recompensation, but there is a marked need for clinical studies investigating novel biomarkers with the capability to predict and monitor improvement in liver cirrhosis, with, and without the impact of alcohol.

Between 75% and 80% of patients with liver cirrhosis in Denmark have or have had a harmful use of alcohol. Dependency of alcohol leads to social isolation, risk of unemployment and a decreased compliance in health care (8). Cirrhosis is related to decreased quality of life and affects patients and relatives both emotional and socioeconomically.

Alcohol related liver disease (ArLD) has a major impact on patients' health and lives, and treatment revolves around symptomatic relief and prevention of further complications. There is an unmet need to investigate treatment options that not only relieves complications, but also address the underlying pathways of alcohol related liver disease, also in severe stages of alcohol related cirrhosis (ALC). Previous studies exploring recompensation in ArLD are retrospective and not designed for the exact purpose.

Factors such as BMI, female gender and minor portal hypertension are known to be associated with an increased likelihood of recompensation. Additional factors of genetic activation and molecular biomarkers from the proteome and lipidome have only attracted minor attention, and the impact of treating the drivers of decompensation, portal hypertension and alcohol use, and their impact on the natural cause of disease, have not been addressed.

The Gastro Unit, Amager-Hvidovre Hospital (AHH) has a record area of 550,000 citizens South and West of Copenhagen. The Gastro Unit is the largest in Denmark, with app. 90 admissions daily. 140 people is diagnosed with liver cirrhosis yearly in our department, either by referral from general practice or by debut of disease during hospital admission. From November 2019 to March 2022, 357 patients were evaluated for liver cirrhosis in the Gastro Unit. 20 % of these died within twelve months. 75% had alcohol use as the primary cause of liver cirrhosis.

Novel molecular technologies and risk prediction The molecular pathophysiology of ArLD is incompletely understood. Characterization of the proteome dynamics across the spectrum of ALD could provide new insights into disease mechanisms of both progression and remission of disease. Recent advances in MS-based proteomics have greatly extended its impact in biomedical and clinical research. It enables the identification and quantification of thousands of proteins, making it suitable for studying disease mechanisms and identification of biomarkers. Prior studies have assessed the proteome in metabolic dysfunction-associated steatotic liver disease (MASH) and alcohol-related fibrosis, and proteomic profiles showed a strong association to severity of liver disease. Studies with consecutive follow-up in the severe stages of ALC are still missing.

MS-based proteomics may identify biomarkers of predictive value in the clinic especially in the prospect of remission of disease. Linkage to clinical data and outcomes may support the use of proteomic biomarkers in the prediction and monitoring of remission in AH and recompensation in ALC.

Several markers of inflammation and cytokines are involved in driving decompensation and has the potential to predict the risk of early death. It is unknown whether such markers can predict remission and recompensation in ALC and AH. Prior studies have assessed relations between inflammation and mortality, but prospective studies investigating the associations between biomarkers of metabolism and prognosis, monitoring and efficacy og treatment in in ALC are missing.

Transcriptomics and gene activation in progression and remission of liver disease The molecular and cellular complexity of the hepatic microenvironment remains a key obstacle hindering the development of potential treatments. Prior studies in RNA sequencing are small and with-out follow-up.

With advances in gene chips and high-throughput sequencing, several prognostic gene signatures have been established to predict overall survival in liver cirrhosis.

Recent single cell RNA sequencing and bulk RNA sequencing studies have shown that specific mesenchymal, endothelial, and monocyte lineages are enriched in cirrhotic livers.

Whole tissue (bulk) RNA sequencing provides an average readout of the RNA content of a sample, which represents mixed RNA signals from the different cells present within the tissue and is thus significantly influenced by cell type prevalence. Compared to single cell RNA sequencing (scRNA-seq), bulk RNA sequencing cannot be used to study rare cell populations, or specific pathogenic cell subpopulations, but it does provide insight into patterns of pathogenic gene transcription and cellular dysfunction, especially when linked to clinical phenotype and when compared to a scRNA- seq library of liver tissue.

No studies have previously compared changes in the transcriptome after removal of the toxic agents causing liver damage.

In ALC, there is an unmet need to investigate treatment options that address the underlying pathways of ArLD, also in severe stages of cirrhosis. Induction of recompensation will prolong both survival and 'admission free' daily life of patients with ALC.

Objectives The overall objective of the present study is to investigate the molecular profile and pathways in persons with ALD to support personalized monitoring and follow-up in liver cirrhosis.

Hypothesis The prognosis of ALC varies depending on continuous or ceased alcohol intake. Alcohol may influence survival and recompensation in ALC. Alcohol may influence the molecular profile of each person with ALC and hence impact hospital admissions, readmissions and progression of liver cirrhosis.

Better knowledge of the molecular profile of persons with ALC will, in combination with clinical features of the patient's health and physical performance, enable us to plan and administer actions of personalized treatment, monitoring and follow-up of people with ALC.

A deeper insight into the molecular mechanisms of the liver driving progression and remission of cirrhosis will -in combination with clinical data- support our ability to predict outcomes in cirrhosis, facilitate personalized monitoring and follow-up and support the right and timely treatment for the right patient. The findings may also support development of novel molecular drug targets for treatment and prevention of cirrhosis in the future.

Methods The study is an incidence cohort in which patients will be followed from diagnosis to death or withdrawal from the cohort. We will seek to include patients consecutively within three months of diagnosis. The results will be reported after STROBE guidelines.

Study subjects All persons with an initial referral to investigation for- and diagnosis of alcohol related liver cirrhosis in the Gastro Unit, and all patients with a debut of alcohol related liver cirrhosis during admission regardless of the reason for admission, are eligible for inclusion.

This study does not compromise diagnostics or treatment of cirrhosis or comorbidities, and inclusion into interventional studies during the prospective follow-up is possible.

Recruitment All patients with a debut of liver cirrhosis suspected to be related to use of alcohol, and irrespective of time and circumstances of diagnosis, comorbidities and severity of disease will be offered inclusion in the cohort. All participants will be engaged by either the physician or nurse providing standard of care. All participants will be informed in writing as well as orally by study investigators and project nurses.

Alcohol cessation intervention and standard of care All patients with ALC treated in the Gastro Unit, AHH, and therefore all participants in this study will be offered the standard of care treatment. This includes investigations with standard biochemistry, ultrasound, fibroscan, CT-scan and endoscopy, as well as nutritional supplements, medical treatment for cirrhosis and complications, and comorbidities.

The alcohol cessation intervention will be offered as standard of care treatment to all patients with ALC. The intervention includes medical treatment of withdrawal symptoms and craving, and support to referral to municipal offers of alcohol treatment. Furthermore, with the aim of facilitating alcohol cessation and supporting further alcohol treatment in the primary sector, the patients will be offered Motivational Interviewing (MI) as part of their treatment.

The patients and possible caregivers will be invited to three MI sessions conducted by specialized nurses in the Liver Clinic within the first three months after diagnosis.

Data from patient journals In this study we will retrieve information from the patient journal after written consent is provided.

Data retrieved from patient journals prior to obtaining consent is limited to the diagnosis of ALC, time of the diagnosis, and the cause of hospital admission or referral that led to diagnosis of ArLD. Biometrical data obtained before written consent to participation will not be retrieved for the study. This data may be collected from a period of zero to thirty days prior to inclusion and will be passed on to clinician investigators, and study personnel.

Data and personal information are registered and monitored after current legislation, The Data Protection Act, and as stated by the General Data protection Regulation.

Genetic analyses DNA will be extracted from blood cells, whole blood and from stool from the participants. The DNA will be stored at -80C, until further analysis. Genotyping will be performed with a GWAS-chip (i.e. targeted genomic mapping) using Illumina Exomechip enriched for protein-changing, large-effect variants. Ultra-rare variants (<1/1000) will not be captured. Results from genetic analyses combined with clinical data may identify genes associated with mortality, survival and severity of disease in a 'risk profiling' context. Genomic analysis comprises common variants and polygenic risk score profiling on common variants. Whole genome sequencing will not be performed.

Genetic analyses on bacterial DNA from stool will be used for comparative analyses of the interplay between intestinal dysfunction and liver cirrhosis.

Transcriptomics, metabolomics and proteomics For identification of novel potential markers involved in development, progression and remission of ALC, transcriptomics, metabolomics and proteomics will be performed on liver tissue and blood. Analyses will evaluate expression levels and cellular localization of possible biomarkers including receptor and ligands as well as downstream signaling molecules. The applied techniques are described below. Together with clinical data, results will improve understanding of possible drivers for remission and progression of ArLD.

The field of discovery omics tenchnologies is rapidly evolving, and methods may be subject to adaptations to secure quality, relevance, and the best prizes for the analysis.

Proteomics analysis Analysis of plasma samples ensures a high success rate and repeated sampling over time is easily tolerated by patients. Snap-frozen liver biopsies will be collected at baseline and at 12 months for analysis. Preparation of samples and liquid chromatography and mass spectrometry (LC/MS) analysis will follow technologies previously described from Torben Hansen and Center for Basic Metabolic Research (CBMR), Copenhagen University. In single-shot plasma proteome analysis, the peptide mixture is eluted Evosep One LC system (Evosep Biosystems) coupled online to an Orbitrap Exploris 480 mass spectrometer.

Lipidomics analyses:

Analysis is performed according to state-of-the-art existing procedures and modified to apply the best available technology.

After plasma preparation, chromatographic separation is performed on Waters Acquity BEH C18 column (1.7μm X 2.1mm X 100 mm) using the gradient of two standard mobile phases (mobile phase A contains water, 0.1% formic acid and 10 ml 1M ammonium acetate, mobile phase B composes isopropanol and acetonitrile (1:1) with the same addition of formic acid and ammonium acetate).

The Mass spectrometry identification of compounds is targeted based on a pre-made library of target metabolites in plasma.

Based on the results from the lipidomics analyses, we will select a panel of diagnostic markers, which will most efficiently describe the speed of the disease progression. For the selected biomarkers we will develop an absolute quantitative method, based on LC-MS-MS (triple quadrupole MS in MRM mode) methodology, using commercially available standard compounds, including stable isotope labelled compounds as internal standards. The method will be validated according to standardized protocols. In the case of successful results, we will be able to set concentration limits of panel biomarkers for prediction of slow, medium, and fast disease progression, as well in the long-term make the method ready to transfer into clinical laboratories and personalized medicine.

The biological analysis and data management of proteomics and lipidomics will take place at the CBMR.

Transcriptomomics analyses Analyses and biostatistics will be performed at Center for Basic Metabolic Research.

Bulk RNA sequencing provides a tissue-wide transcription landscape and allows for deep investigation into the transcriptome, but it does not distinguish between individual cells. To identify genes that play an important role in the progression or recompensation of AH, we will compare datasets from bulk RNA sequencing in AH to already established datasets from single cell RNS sequencing of the liver.

Based on genes that are simultaneously suggested by bulk-RNA in our samples and scRNAseq, we can explore the key transcriptional regulators in ALC.

We will make use of this resource to computationally deconvolute the bulk transcriptome data of the liver biopsies to estimate the relative abundance of each cell type of the liver (hepatocyte, hepatic stellate cells, liver sinusoidal epithelial cells, etc.) in each patient. Possible disease regulators of both progression and recompensation will be assessed.

Research biobank A biobank will be established for the study. The biobank will contain blood collected at baseline, three months, 1 and 3 years, and liver tissue and stool collected at baseline and after 1 year. At each time point, 15 ml of blood and 3 gram of stool is collected. At baseline and after 1 year 0,2 gram of liver tissue will be collected. If a participant has ascites and needs paracentesis, a subcutaneous fat biopsy will be taken from the incision spot on the abdomen.

Surplus material from the study will be transferred to a biobank for future research.

Perspectives The study will contribute to a better characterization of advanced liver disease related to alcohol and contribute to an improved future organization of treatment- and rehabilitation offers to patients with liver disease. thorough characterization and consecutive inclusion will enhance our understanding on the incidence, prevalence and impact of ALC in the population, as well as the utilization of health care resources allocated to its treatment.

A deeper insight into the molecular mechanisms of liver progression and remission will, in combination with clinical data, support our ability to predict outcomes in cirrhosis, facilitate personalized monitoring aiming at providing the right treatment for the right patient at the right time.

The prospective cohort study will further contribute to the identification of previously unidentified risk factors significant for survival and the use of health care services; and thereby form the basis of implementing changes in health practices that offer both economic and medical benefits. Additionally, the study may uncover new areas for interventional research with clinically relevant endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Clinical suspicion of cirrhosis related to use of alcohol, supported by biochemistry and ultrasound or other imaging techniques.
* Informed written consent.

Exclusion Criteria:

* The diagnosis of ALC is questioned with reasonable doubt.
* Withdrawal of informed consent or no informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2024-12-22 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Survival | 12 months
  Mortality

SECONDARY OUTCOMES:
Recompensation | 12 months
  Rate of patients free from decompensation
Alcohol use | 12 months
  Change in use of alcohol by 30 days timeline follow-back (total use of alcohol in 30 days)
Clinical improvement | 12 months
  Change in MELD (Creatinine, INR, bilirubin)
Alcohol use | 12 months
  Change in use of alcohol by 30 days timeline follow-back (total days with alcohol use in 30 days)

OTHER OUTCOMES:
Lipid profile | 12 months
  Changes in lipidomic profile in plasma
Proteomic profile | 12 months
  Changes in proteomic profile in plasma
Metabolic changes in the liver | 12 months
  Changes in metabolic profile in the liver over time

CONTACTS AND LOCATIONS:
Overall Officials: Nina Kimer, MD, PhD, Principal Investigator — Gastroenheden, Hvidovre Hospital
Locations (1):
- Copenhagen University Hospital Hvidovre, Hvidovre, Capital Region, Denmark